CLINICAL TRIAL: NCT02937350
Title: Clearance of 25-hydroxyvitamin D in Chronic Kidney Disease
Acronym: CLEAR
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Ian deBoer, Professor, Medicine/Nephrology, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY00009578; R01DK099199 (NIH)
Record Dates: First submitted 2016-10-14; First posted 2016-10-18 (Estimated); Results first posted 2021-09-01 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Chronic Kidney Disease
Keywords: chronic kidney disease; vitamin d catabolism
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Study Population (Experimental): D6-25-hydroxyvitamin D3
  Interventions: Drug: D6-25-hydroxyvitamin D3

INTERVENTIONS:
Drug: D6-25-hydroxyvitamin D3 — Intravenous administration of a deuterium-labeled 25(OH)D3 to evaluate the metabolic clearance of 25(OH)D3
  Other Names: stable isotope deuterium-labeled 25(OH)D3

SUMMARY:
The goal of this study is to better understand vitamin D catabolism and how it is affected by CKD and race.

DETAILED DESCRIPTION:
Specifically, the study team will evaluate the metabolic clearance of 25-hydroxyvitamin D3 in individuals with varying degrees of CKD and among participants who self-report race as Caucasian, African American or African. The long-term goal of this work is to enhance the clinical evaluation and treatment of impaired vitamin D metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Self-reported race Caucasian, African American, or African
* Serum total 25(OH)D 10-50 ng/mL
* Estimated GFR:

  * 60 mL/min/1.73m2 (N=40) 15-45 mL/min/1.73m2 (N=40) <15 mL/min/1.73m2, treated with hemodialysis (N=40)

Exclusion Criteria:

* Primary hyperparathyroidism
* Gastric bypass
* Tuberculosis or sarcoidosis
* Current pregnancy
* Child-Pugh Class B or C cirrhosis (i.e. cirrhosis with ascites, hepatic encephalopathy, bilirubin >=2 mg/dL, serum albumin <=3.5 g/dL, or PT >= 4 seconds)
* Use of vitamin D3, or vitamin D2 supplements exceeding a mean daily dose of 400 IU, within 3 months (wash-out allowed)
* Use of 1,25(OH)2D3 or an analogue, calcimimetics, or medications known to induce CYP24A1 within 4 weeks (wash-out allowed)
* Serum calcium > 10.1 mg/dL
* Hemoglobin < 10 g/dL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-07-08 (Actual); Study Completion 2021-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian de Boer, MD, MS, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Best CM, Thummel KE, Hsu S, Lin Y, Zelnick LR, Kestenbaum B, Kushnir MM, de Boer IH, Hoofnagle AN. The plasma free fraction of 25-hydroxyvitamin D3 is not strongly associated with 25-hydroxyvitamin D3 clearance in kidney disease patients and controls. J Steroid Biochem Mol Biol. 2023 Feb;226:106206. doi: 10.1016/j.jsbmb.2022.106206. Epub 2022 Oct 28. PMID 36404469
- [Derived] Hsu S, Zelnick LR, Lin YS, Best CM, Kestenbaum B, Thummel KE, Rose LM, Hoofnagle AN, de Boer IH. Differences in 25-Hydroxyvitamin D Clearance by eGFR and Race: A Pharmacokinetic Study. J Am Soc Nephrol. 2021 Jan;32(1):188-198. doi: 10.1681/ASN.2020050625. Epub 2020 Oct 28. PMID 33115916

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Controls: Healthy controls defined as normal eGFR (>60 ml/min per 1.73m2)
- CKD Group: CKD group defined as those with eGFR <60ml/min per 1.73 m2)
- Kidney Failure Group: Kidney failure group defined as those with ESKD treated with dialysis
Period: Overall Study
Arm/Group | Healthy Controls | CKD Group | Kidney Failure Group
Started | 43 | 25 | 20
Completed | 43 | 24 | 20
Not Completed | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Controls | CKD Group | Kidney Failure Group | Total
Number analyzed (Participants) | 43 | 24 | 20 | 87
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (10) | 67 (11) | 58 (9) | 64 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 8 | 4 | 36
  Male | 19 | 16 | 16 | 51
Race (NIH/OMB) [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 0 | 0 | 0 | 0
  Race: Asian | 0 | 0 | 0 | 0
  Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Race: Black or African American | 12 | 8 | 6 | 26
  Race: White | 31 | 16 | 14 | 61
  Race: More than one race | 0 | 0 | 0 | 0
  Race: Unknown or Not Reported | 0 | 0 | 0 | 0
Vitamin-D3 Supplement Use [Number; unit: participants] | 6 | 1 | 1 | 8

OUTCOME MEASURES:

1. Primary Outcome: Metabolic Clearance of D6-25(OH)D3
Description: Metabolic clearance is calculated as the administered dose of 25(OH)D3 divided by the area under the plasma concentration-time curve (AUC). AUC is calculated using the linear trapezoidal method. Concentration was measured at 5 minutes, 4 hours, and at 1, 4, 7, 14, 21, 28, 42, and 56 days post administration.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: milliliter per day (ml/d)
Arm/Group | Healthy Controls | CKD Group | Kidney Failure Group
Number analyzed (Participants) | 43 | 24 | 20
milliliter per day (ml/d) | 360 (108) | 313 (86) | 263 (163)

2. Secondary Outcome: AUC of D6-25(OH)D3
Description: AUC is calculated using the linear trapezoidal method. Concentration was measured at 5 minutes, 4 hours, and at 1, 4, 7, 14, 21, 28, 42, and 56 days post administration.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: nanograms x day/mL (ngxd/mL)
Arm/Group | Healthy Controls | CKD Group | Kidney Failure Group
Number analyzed (Participants) | 43 | 24 | 20
nanograms x day/mL (ngxd/mL) | 59.8 (10.2) | 68.7 (10.2) | 76.6 (12.0)

3. Secondary Outcome: Terminal Half-life of D6-25(OH)D3
Description: Terminal half-life is equal to ln2/k, where k is the slope of the terminal regression line estimated using ≥3 plasma concentrations. Concentration was measured at 5 minutes, 4 hours, and at 1, 4, 7, 14, 21, 28, 42, and 56 days post administration.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: days (d)
Arm/Group | Healthy Controls | CKD Group | Kidney Failure Group
Number analyzed (Participants) | 43 | 24 | 20
days (d) | 21.9 (5.7) | 25.5 (6.5) | 35.6 (8.1)

4. Secondary Outcome: Volume of Distribution of D6-25(OH)D3
Description: Volume of distribution in the central compartment is calculated as dose/C0, where dose is the administered dose of 25(OH)D3 and C0 is the initial (estimated) concentration of drug in plasma. Concentration was measured at 5 minutes, 4 hours, and at 1, 4, 7, 14, 21, 28, 42, and 56 days post administration.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: Liters (L)
Arm/Group | Healthy Controls | CKD Group | Kidney Failure Group
Number analyzed (Participants) | 43 | 24 | 20
Liters (L) | 11.0 (2.9) | 11.1 (2.8) | 12.5 (4.0)

5. Other Pre Specified Outcome: Metabolic Formation Clearance of D6-25(OH)D3 Metabolites.
Description: Metabolic formation clearance is calculated as the daughter metabolite plasma AUC divided by the AUC of D6-25(OH)D3 (metabolite/parent AUC ratio). AUC is calculated using the linear trapezoidal method. Concentration was measured at 5 minutes, 4 hours, and at 1, 4, 7, 14, 21, 28, 42, and 56 days post administration.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Healthy Controls | CKD Group | Kidney Failure Group
Number analyzed (Participants) | 43 | 24 | 20
ratio | 0.12 (0.04) | 0.08 (0.03) | 0.03 (0.03)

6. Other Pre Specified Outcome: Change in the Serum Concentration of Calcium
Description: Change in the serum concentration of calcium from baseline to 7 days after 25(OH)D3 administration
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: milligrams/deciliter (mg/dl)
Arm/Group | Healthy Controls | CKD Group | Kidney Failure Group
Number analyzed (Participants) | 43 | 24 | 20
milligrams/deciliter (mg/dl) | 0.42 (1.75) | 0.16 (0.26) | -0.27 (0.48)

7. Other Pre Specified Outcome: Change in the Serum Concentration of Creatinine
Description: Change in the serum concentration of creatinine from baseline to 7 days after 25(OH)D3 administration
Time Frame: Baseline, 7 days
Measure: Mean (Standard Deviation); unit: milligrams/deciliter (mg/dl)
Arm/Group | Healthy Controls | CKD Group | Kidney Failure Group
Number analyzed (Participants) | 43 | 24 | 20
milligrams/deciliter (mg/dl) | 0.04 (0.09) | -0.05 (0.27) | 2.81 (2.26)

8. Other Pre Specified Outcome: Change in the Serum Concentration of AST
Description: Change in the serum concentration of AST from baseline to 7 days after 25(OH)D3 administration
Time Frame: Baseline, 7 days
Measure: Mean (Standard Deviation); unit: units/Liter (u/L)
Arm/Group | Healthy Controls | CKD Group | Kidney Failure Group
Number analyzed (Participants) | 43 | 24 | 20
units/Liter (u/L) | 0.40 (3.43) | 0.57 (5.98) | 0.10 (5.22)

9. Other Pre Specified Outcome: Change in the Serum Concentration of ALT
Description: Change in the serum concentration of ALT from baseline to 7 days after 25(OH)D3 administration
Time Frame: Baseline, 7 days
Measure: Mean (Standard Deviation); unit: units/Liter (u/L)
Arm/Group | Healthy Controls | CKD Group | Kidney Failure Group
Number analyzed (Participants) | 43 | 24 | 20
units/Liter (u/L) | 0.16 (3.71) | 1.52 (6.92) | 0.45 (3.66)

ADVERSE EVENTS:
Time Frame: 8 weeks
Description: Everyone had the same treatment, so it was more appropriate to summarize AEs for the whole group. Adverse events were not collected separately per arm.
Groups:
- All Participants: All participants (N=87)
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/87
Serious Adverse Events (participants affected / at risk) | 1/87
Other Adverse Events (participants affected / at risk) | 16/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=87)
Deep vein thrombosis (Blood and lymphatic system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=87)
Pain or sensation in arm during infusion (General disorders) | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-10): https://cdn.clinicaltrials.gov/large-docs/50/NCT02937350/Prot_SAP_000.pdf